CLINICAL TRIAL: NCT04806282
Title: Deep Phenotyping of Hearing Instability Disorders: Cohort Establishment, Biomarker Identification, Development of Novel Phenotyping Measures, and Discovery of Therapeutic Targets
Status: Suspended | Type: Observational
Why Stopped: Pause in study enrollment due to PI departure from NIH. IC leadership and the new PI have initiated a pause in the enrollment of new participants to assess the the study s operational capacity.
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000141; 000141-DC
Record Dates: First submitted 2021-03-18; First posted 2021-03-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12-04

CONDITIONS: Meniere's Disease; Enlarged Vestibular Aqueduct Syndrome; Autoimmune Inner Ear Disease
Keywords: Biomarkers; immunoprofiling; Auditory
MeSH Terms: conditions — Meniere Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/All Patients: Documented hearing instability

SUMMARY:
Background:

Disorders of hearing instability (HI) are poorly characterized and ineffectively treated. HI can cause fluctuations in hearing thresholds and speech understanding. Researchers want to use a specialized form of magnetic resonance imaging (MRI) and blood tests to learn more about HI.

Objective:

To characterize a cohort of people with HI and to correlate HI with other data, including hearing evaluations, as well as radiologic and immunologic biomarkers of inflammation over time.

Eligibility:

Adults ages 18-80 who have symptoms consistent with possible HI.

Design:

Participants will be screened with a medical and hearing history and medical record review.

Participants will have physical exams. Their head and neck will be examined. They will have blood drawn.

Participants will have hearing tests. They will wear headphones or foam earplugs. They will listen to different tones. They may describe what they hear.

Participants will have balance tests. They will wear goggles as they watch moving lights or while cold or warm air is blown into their ears. They will sit in a spinning chair in a quiet, dark booth. From a reclining position, they will raise their head while clicking sounds are played into their ears.

Participants will have MRIs of the inner ear and brain. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the MRIs, participants will lie on a table that slides in and out of the scanner. Soft padding or a coil will be placed around their head. They will get a contrast agent through an intravenous catheter.

Participation will last up to 15 months.

...

DETAILED DESCRIPTION:
Study Description:

Disorders of hearing instability remain poorly characterized, phenotyped and ineffectively treated, and may result in sudden changes in hearing. These disorders include, but are not limited to, sudden sensorineural hearing loss (SSNHL) as well as hearing fluctuation, including, but not limited to, autoimmune inner ear disease (AIED), Meniere s disease (MD) and enlarged vestibular aqueduct syndrome (EVAS). While this group of disorders is likely to be clinically and etiologically heterogeneous, a common feature is fluctuation of hearing thresholds and speech understanding as measured by word recognition scores (WRS). This protocol seeks to ascertain a cohort of patients with hearing fluctuation to correlate these main phenotypic features with other phenomic data including audiometric indicators of endolymphatic hydrops as well as radiologic and immunologic biomarkers of inflammation over time. The overall hypothesis is that phenomic data will enable stratification of the phenotype of patients with hearing instability disorders. Healthy volunteers will be recruited to establish the normative range of endolymph and perilymph on contrast-enhanced delayed FLAIR MRI to allow for quantitative computational analysis of contrastenhanced delayed FLAIR MRI images.

Objectives:

Primary objective: To develop a cohort of patients with hearing instability (HI).

Secondary objectives:

1. To correlate evidence of HI with changes in phase-shift distortion product otoacoustic emissions (DPOAEs).
2. To compare phase-shift DPOAEs to existing measures of auditory function including word recognition score (WRS), standard DPOAEs, and electrocochleography (ECochG) over time.
3. To compare phase-shift DPOAEs to vestibular measures including cervical and ocular vestibular evoked myogenic potentials (VEMPs) over time.
4. To correlate auditory and vestibular indicators of hearing instability and endolymphatic hydrops (EH) on MRI with quantitative differences in immunologic markers of inflammation over time.
5. Establish the normative range of endolymph and perilymph volume on contrast-enhanced delayed FLAIR MRI to allow for quantitative computational analysis of contrast-enhanced delayed FLAIR MRI images

Exploratory objective:

1. To stratify patients with hearing instability (HI) by differences in cytokine levels, which will inform the identification of clinical subtypes of HI and potentially identify therapeutic targets for future treatment with targeted agents.
2. To perform transcriptional and immunoprofiling of PBMCs at time points associated with hearing fluctuation from phenotyped patient cohorts.

Endpoints:

Primary Endpoint: Identification of phenomic features associated with HI.

Secondary Endpoint:

(1) Identification of a variety of phenomic features of patients with HI that allow assignment to clinical subdivisions.

Exploratory Endpoints

1. Identification of potential targets for therapeutics based on longitudinal immune/transcriptional profiling of patients with hearing instability.
2. Identification of subtype-specific immune cell distributions
3. Identification of immune profiles as well as immune cell transcriptional profiles related to hearing fluctuation

ELIGIBILITY:
* NCLUSION CRITERIA:

Affected Adults

In order to be eligible to participate in this study as a subject with HI, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent.
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. All genders, aged 18-80 years

   Diagnosed with hearing instability, defined as documented hearing instability on serial audiometry with sensorineural hearing loss (SNHL) greater than 30 dB HL at one or more frequencies on at least one hearing test. Inclusion will require documentation of clinically significant change in hearing (either worsening or improvement) between at least 2 hearing tests or documentation of a sudden change in hearing. Clinically significant change in hearing will be defined by a change of10 dB at any three frequencies, 15 dB at any two frequencies, or at least 20 dB at one frequency. A sudden change in hearing will be defined as at least a 30 dB difference at 3 consecutive frequencies in the affected ear as compared to the contralateral ear.
4. No air-bone gaps in excess of 10 dB for 500-4000 Hz indicative of conductive HL in at least 1 ear.
5. For females of reproductive potential: Negative pregnancy test at start of study

Unaffected Adults

In order to be eligible to participate in this study as a healthy volunteer, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent.
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. All genders, aged 18-80 years
4. No air-bone gaps in excess of 10 dB for 500-4000Hz indicative of conductive HL in at least one ear.
5. Normal middle ear function as indicated by normal 226 Hz tympanograms bilaterally, defined as middle ear pressure between plus minus 100 decaPascals, and peak compensated static compliance between 0.3-1.8 milliliters
6. For females of reproductive potential: Negative pregnancy test at start of study

EXCLUSION CRITERIA:

Affected and unaffected individuals who meet any of the following criteria will be excluded from participation in this study:

1. Presence of non-MRI compatible devices (cardiac pacemaker, meta<specific devices (e.g., cardiac pacemaker)
2. Pregnancy or lactation
3. Known allergic reactions to gadolinium
4. Febrile illness within 2 weeks that could affect immune profiling*
5. Evidence of active outer or middle ear disease or anomaly (e.g. otitis media, stenotic ear canal, otorrhea)
6. History of chronic, as defined by fluid in the middle ear for more than 4 months, or recurrent otitis media, as defined by more than 4 episodes of acute otitis media in one year.
7. Current PE tubes
8. Bilateral profound (Pure tone average (PTA) > 90 dB HL) sensorineural hearing loss
9. History or diagnosis of a central nervous system disorder, including but not limited to:

   1. Intracranial tumors
   2. Cerebrovascular disease
   3. Degenerative CNS disorder
   4. CNS trauma
   5. Encephalitis
   6. Meningitis
10. Unable to discontinue medications that can interfere with vestibular test results for the 48 hours immediately preceding a vestibular study session. These include any and all anti-dizziness medications (such as Antivert), alcohol, caffeine, prescription pain medications (such as Percocet), prescription headache medications (such as Imitrex), sleeping pills (such as Ambien), anti-seizure medications (such as Topamax), and/or antihistamines (such as Benadryl).
11. Current diagnosis from the Diagnostic and Statistical Manual of Mental Disorders (DSM IV) of schizophrenia, bipolar disorder, or psychosis.
12. Unstable intercurrent illness that in the judgment of the PI could prevent or confound collection of data.

Prospective study subjects who are cognitively impaired and lack consent capacity, will not be enrolled.

*Participants suspected of having COVID-19 will be moved to the designated COVID-19 unit and tested for SARS CoV-2 and Respiratory Pathogen Panel per guidance from NIH CC Clinical Practice Safety Guidelines. Possible COVID-19 infections identified by phone screen will not be eligible for study protocol until infection resolved.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll up to a total of 150 patients with HI. The enrollment target is between 10-30 patients per clinical subtype for at least 2 clinical subtypes of HI (i.e., without or with EH, without or with significant immune cell, cytokine or FLAIR positivity). 20 cytokines/chemokines in patients with Meniere s disease that revealed statistically higher levels of IL-1Beta compared to healthy controls (Flook et al., 2019), a sample size of 40-50 patients would be required for 80% power to detect an immune subtype associated with IL-1Beta.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Phenomic features | Day 90, 180, 270, 360, and 450, respectively +/- 14 days
  To identify phenotype features associated with hearing fluctuation

SECONDARY OUTCOMES:
Subdivisions of phenomic features | Day 90, 180, 270, 360, and 450, respectively +/- 14 days
  To Identify a variety of phenomic features of patients with HI that allow assignment to clinical subdivisions.

CONTACTS AND LOCATIONS:
Overall Officials: Ronna P Hertzano, M.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Telischi J, Strepay D, Li B, Chisholm J, Cheng H, Brewer C, Hsu LY, Butman J, Hoa M. MRI-based measurement of inner ear fluids reveals increased endolymph volume variability in patients with endolymphatic hydrops and hearing instability. Sci Rep. 2025 Jul 2;15(1):22560. doi: 10.1038/s41598-025-06083-w. PMID 40596438
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000141-DC.html